CLINICAL TRIAL: NCT03301961
Title: The Clinical Applications of Multiplex Analysis of Circulating Tumor DNA Biomarkers in Lung Cancer Patients
Brief Title: Multiplex Analysis of Circulating Tumor DNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Jun Wang, Chief，Thoracic Surgery Service, Peking University People's Hospital
Other Study IDs: PTHO1701
Record Dates: First submitted 2017-09-30; First posted 2017-10-04 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Carcinoma; Non-small-cell Lung Cancer; Lung Neoplasm
Keywords: Circulating Tumor DNA; Early diagnosis; Surveillance; Methylation; Somatic mutation
MeSH Terms: conditions — Carcinoma; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — A series of lung cancer patients plasma before and after surgery
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Lung cancer is the leading cause of cancer-related death in China. This study will explore the applications of multiplex analysis of circulating tumor DNA biomarkers for diagnosis and surveillance of lung cancer patients

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) constitutes about 85% of all newly diagnosed cases of lung cancer and continues to be the leading cause of cancer-related deaths worldwide.Early diagnosis and monitoring tumor recurrence after surgery are still far from satisfying.

Circulating tumor DNA(ctDNA) detection has been proved to be feasible in early stage NSCLC in previous studies.Both genomic mutation and methylation a promising biomarker.Therefore,this study will perform multiplex detection of ctDNA,analysing mutations, methylation and other biomarkers,focusing on the early diagnosis and postoperative surveillance for NSCLC patients.

ELIGIBILITY:
Inclusion Criteria:

1. Sign informed consent and consent to participate in this study;
2. Found small nodules in pulmonary by CT and prepare for surgery;

Exclusion Criteria:

1. Malignant tumor history within the past 5 years;
2. Receiving chemotherapy, radiotherapy or targeted therapy before surgery;
3. No matching tissue or blood samplesUnqualified blood samples
4. Lesion is pure ground glass opacity.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patient are found nodules in pulmonary and prepare for surgery
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2019-04-11 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of multiplex peripheral blood ctDNA biomarkers in the diagnosis of non-small cell lung cancer | 12 months

SECONDARY OUTCOMES:
Comparing the sensitivity and specificity of each peripheral blood biomarkers for the diagnosis of non-small cell lung cancer | 12 months
The sensitivity and specificity of multiplex peripheral blood ctDNA biomarkers for tumor relapse detection | 36 months
Lead time of tumor relapse detection by multiplex ctDNA biomarkers than radiographic approaches | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Kezhong Chen, MD, Study Director — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, Beijing Municipality, China